CLINICAL TRIAL: NCT02424578
Title: A Phase IIA, Open-Label, Safety and Pharmacokinetic Study of Diclofenac Capsules in Pediatric Subjects 6 to <17 Years of Age With Mild to Moderate Acute Postoperative Pain Following Elective Surgery
Brief Title: Study of Diclofenac Capsules to Treat Pain Following Surgery in Children Ages 6 to <17 Years of Age
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Iroko Pharmaceuticals, LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DIC2-14-08
Record Dates: First submitted 2015-04-20; First posted 2015-04-23 (Estimated); Results first posted 2017-07-13 (Actual); Last update posted 2017-07-13 (Actual); Status verified 2017-06

CONDITIONS: Pain, Postoperative
MeSH Terms: conditions — Pain, Postoperative | interventions — Diclofenac

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Diclofenac Capsules low dose (Experimental): Diclofenac Capsules low dose three times daily for up to three days
  Interventions: Drug: Diclofenac Capsules low dose
- Diclofenac Capsules high dose (Experimental): Diclofenac Capsules high dose three times daily for up to three days
  Interventions: Drug: Diclofenac Capsules high dose

INTERVENTIONS:
Drug: Diclofenac Capsules low dose
  Arms: Diclofenac Capsules low dose
Drug: Diclofenac Capsules high dose
  Arms: Diclofenac Capsules high dose

SUMMARY:
The purposes of this study are to evaluate the safety and tolerability and to model the single-dose pharmacokinetic profile of diclofenac capsules low dose and high dose in children ages 6 to <17 years experiencing mild to moderate acute postoperative pain.

ELIGIBILITY:
Inclusion Criteria:

* Body weight ≥18 kilograms.
* Mild to moderate acute pain requiring treatment with analgesic medication.
* Willing to have blood samples taken for PK sampling using an indwelling catheter.
* Must be able to swallow capsules and can tolerate oral medication.
* For females: is not of reproductive potential (defined as premenarchal) or is practicing an acceptable method of birth control

Exclusion Criteria:

* Severe acute pain
* Chronic analgesic or glucocorticoid use for any condition within 6 months before dosing with study drug.
* Emergency surgery
* History of allergic reaction, hypersensitivity, or clinically significant intolerance to diclofenac, aspirin, codeine, acetaminophen, or any NSAID
* History of peptic ulcer disease or a GI event (eg, perforation, obstruction, or bleed) within 6 months before screening
* Current use of any medication that may cause a clinically significant drug interaction when co-administered with diclofenac
* Current use of any medication that might affect the pharmacokinetics of diclofenac
* History of bleeding disorders .
* Developmental delay or behavioral problems that would make it difficult to assess pain.
* Impaired liver function
* Clinically significant renal or cardiovascular disease
* Any medical condition that compromises ability to swallow, absorb, metabolize, or excrete the study drug
* Previously received any investigational product or device within 30 days before Screening or scheduled to receive an investigational device or another investigational drug (other than that in this study) during the course of this study.
* Previous participation in this clinical study or currently taking diclofenac.

Ages: 6 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2015-05; Primary Completion 2016-04 (Actual); Study Completion 2016-04-19 (Actual)

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Sheffield, Alabama
  - Little Rock, Arkansas
  - Durham, North Carolina
  - Oklahoma City, Oklahoma
  - Philadelphia, Pennsylvania

RESULTS

PARTICIPANT FLOW:
Groups:
- Diclofenac Capsules Low Dose: Diclofenac Capsules low dose three times daily for up to three days
  Diclofenac Capsules low dose
- Diclofenac Capsules High Dose: Diclofenac Capsules high dose three times daily for up to three days
  Diclofenac Capsules high dose
Period: Overall Study
Arm/Group | Diclofenac Capsules Low Dose | Diclofenac Capsules High Dose
Started | 15 | 15
Completed | 15 | 14
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Population: Safety Population (all subjects receiving at least one dose of study medication)
Groups:
- Total: Total of all reporting groups
Arm/Group | Diclofenac Capsules Low Dose | Diclofenac Capsules High Dose | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 15 | 15 | 30
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 9.0 (1.69) | 14.1 (1.51) | 11.6 (3.05)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 6 | 17
  Male | 4 | 9 | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 15 | 15 | 30
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 2 | 7
  White | 9 | 11 | 20
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 1 | 1 | 2
Weight [Mean (Standard Deviation); unit: kg] | 40.20 (16.628) | 74.44 (18.974) | 57.34 (24.693)
Weight Group [Count of Participants; unit: Participants]
  >/=18 to <35 kg | 7 | 0 | 7
  >/=35 kg | 8 | 15 | 23

OUTCOME MEASURES:

1. Primary Outcome: Plasma Concentration of Diclofenac
Description: The estimated typical value for clearance (tvCl) following a single diclofenac dose based on population pharmacokinetic (PopPK) modeling using sparse plasma concentration data in pediatric subjects.
Time Frame: 0-6 hours after first dose of diclofenac
Population: Pharmacokinetic (PK) population. Defined as all subjects who received at least one dose of study drug and had at least one quantifiable plasma diclofenac concentration after dosing.
Measure: Mean (Standard Error); unit: mL/hr
Arm/Group | Diclofenac Capsules Low Dose | Diclofenac Capsules High Dose
Number analyzed (Participants) | 15 | 15
mL/hr | 29647.9 (3710.526) | 35131.0 (5660.83)

2. Secondary Outcome: Safety of Diclofenac Capsules Low Dose and High Dose as Assessed by the Incidence of Adverse Events From Baseline to Day 3 or Early Termination
Time Frame: Baseline to Day 3/Early Termination
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse Events (AEs) were collected from the signing of the informed consent document, through the study follow up visit (approximately 1 week after the final dose of diclofenac).
Description: Standard AE definitions were used. AE data were collected using non-leading questioning for subjects who were inpatients, and were collected using a take-home signs and symptoms diary (with parent/guardian assistance) for outpatient subjects. Daily phone calls were made to outpatient subjects to ensure compliance with diary collection procedures.
Arm/Group | Diclofenac Capsules Low Dose | Diclofenac Capsules High Dose
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/15
Serious Adverse Events (participants affected / at risk) | 1/15 | 0/15
Other Adverse Events (participants affected / at risk) | 7/15 | 7/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Diclofenac Capsules Low Dose (N=15) | Diclofenac Capsules High Dose (N=15)
Postoperative abcess (Infections and infestations) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Diclofenac Capsules Low Dose (N=15) | Diclofenac Capsules High Dose (N=15)
Nausea (Gastrointestinal disorders) | 0 (0) | 3 (3)
Vomiting (Gastrointestinal disorders) | 2 (3) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pain (General disorders) | 1 (1) | 0 (0)
Pharyngitis streptococcal (Infections and infestations) | 1 (1) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0)
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less